CLINICAL TRIAL: NCT03405246
Title: Keeping Ideal Cardiovascular Health Family Intervention Trial (KIDFIT)
Brief Title: KIDFIT: Keeping Ideal Cardiovascular Health Family Intervention Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northwestern University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Linda Van Horn, Professor, Northwestern University, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17SFRN33700242
Record Dates: First submitted 2018-01-12; First posted 2018-01-23 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2021-08

CONDITIONS: Childhood Obesity; Weight Gain; Diet Modification
Keywords: Childhood obesity; Weight gain in children; Diet intervention
MeSH Terms: conditions — Pediatric Obesity; Weight Gain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KIDFIT SAFE (Active Comparator): The Control Group will be provided 12 web-based monthly Homestyles Safe Guides about safe home environments for raising children and related material emailed monthly to the moms. KIDFIT Safe web site targets environmentally safe childcare related topics such as use of sun screen, avoidance of choking hazards, pet safety, protection from electrical appliances, etc. KIDFIT Safe participants will attend both baseline and 12 month clinical visits.
  Interventions: Behavioral: KIDFIT SAFE
- KIDFIT HEALTHY (Experimental): The KIDFIT intervention group combines traditional in-person and electronic participant contacts, including two scheduled individual visits with a nutrition coach, coaching calls throughout the year, and monthly group videoconferencing-type sessions. KIDFIT Healthy participants will attend both baseline and 12 month clinical visits.
  Interventions: Behavioral: KIDFIT HEALTHY

INTERVENTIONS:
Behavioral: KIDFIT HEALTHY — KIDFIT Healthy intervention combines traditional in-person and electronic participant contacts.
  Other Names: Intervention Group
  Arms: KIDFIT HEALTHY
Behavioral: KIDFIT SAFE — KIDFIT Safe group will be referred to the KIDFIT Safe website for monthly Homestyles Safe Guides about safe home environments for raising children and related material emailed monthly to the moms.
  Other Names: Control Group
  Arms: KIDFIT SAFE

SUMMARY:
Adverse influences starting in utero may predestine an individual's long- term risk for developing cardiometabolic diseases. The Keeping Ideal CVH (cardiovascular health) Family Intervention Trial (KIDFIT) will test whether preschool-age children, born to overweight/obese (OW/OB (mothers who did or did not experience a diet and lifestyle intervention to reduce GWG: 1) demonstrate more favorable adiposity (body fat %), body mass index percentiles (BMI%), diet quality (DASH diet score), physical activity, and other CVH metrics at baseline according to antenatal intervention status; and 2) respond to an early childhood intervention targeting diet and lifestyle behaviors with improvement in these same adiposity and CVH metrics.

We hypothesize children randomized to the KIDFIT diet and lifestyle intervention group at age 3-5 years, regardless of initial maternal antenatal group assignment, will demonstrate more favorable adiposity changes assessed by anthropometry (body fat %/sum of skinfolds) and a lower cumulative incidence of obesity after the 12-month intervention, as compared with the control group. Additionally, after 12 months of the KIDFIT Intervention, children will have more favorable blood pressure and blood lipids, better diet quality (as measured by the DASH-style diet score), increased physical activity levels, and more optimal sleep duration, without adverse effects on height, compared to the control group

DETAILED DESCRIPTION:
A randomized controlled trial (RCT) is planned among 140 of the MOMFIT offspring, aged 3-5 years old. The KIDFIT Study follows final data collection in the MOMFIT RCT. Moms were randomized to either the MAMA DASH Diet and lifestyle intervention or the "Web-Watcher" enhanced usual care group that received periodic newsletters highlighting publicly available websites and reputable links related to healthy pregnancy. The first MOMFIT baby was born in September 2013 and the last was born in July 2016; the KIDFIT cohort will include children who are ages 3-5 years at the time of randomization. Post-partum, the MAMA DASH Intervention Group received ongoing encouragement for maternal adherence to the DASH Diet and breastfeeding of the child for as long as possible, preferably at least six months. General diet information regarding post-weaning was provided briefly to further encourage maternal adherence to the diet. KIDFIT will randomize children stratified by the original MOMFIT groups to either the DASH Diet and Lifestyle intervention (called KIDFIT-Healthy) or enhanced (websites/apps) Usual Care called KIDFIT-Safe. Children randomized to the intervention group will have a 12 month diet and lifestyle intervention that will implement the DASH kids diet, encourage physical activity, limit screen time, and encourage 10 to 13 hours of sleep. Mother-Child Dyads randomized to the usual care group will be sent monthly guides addressing environmentally safe home settings to raise children and given related resources for healthy family lifestyle habits for their family.

The KIDFIT clinical intervention will develop, implement and test a lifestyle intervention to determine whether (1) children ages 3-5 years, born to overweight/obese (OW/OB) mothers who adhered to an antenatal diet and lifestyle intervention, demonstrate improvements in weight gain trajectories, diet pattern quality, physical activity levels and other ideal cardiovascular health (iCVH) measures compared to children whose OW/OB mothers underwent usual care; (2) lifestyle intervention at ages 3-5 years is associated with improvements in those same measures independent of or additive to maternal intervention; and (3) epigenetic mechanisms and molecular pathways underlying these associations can be differentiated.KIDFIT results will help determine whether antenatal diet and lifestyle interventions and/or early life child-focused diet and lifestyle interventions offer the potential for prevention of obesity, thereby maintaining iCVH earlier and longer.

ELIGIBILITY:
Inclusion Criteria: Because this cohort includes former participants of the MOMFIT study, there are certain pre-existing criteria regarding the health, age, and antenatal BMI (25-40 kg/m2) among the mothers of the KIDFIT children. In addition, eligibility for this study requires willingness of the mother/child dyad:

* to be randomized
* to attend study visits and participate in intervention sessions
* to monitor the child's diet, physical activity, and sleep

Exclusion Criteria:

* planning to move away within 18 months
* child has a medical condition (e.g. fed by gastric tube, wheelchair user) that limits ability or willingness to adhere to diet and activity recommendations (parents will be encouraged to discuss with their pediatrician if there is any question)
* child is already under the care of a nutritionist and mother and/or nutritionist unwilling to collaborate with KIDFIT Dietitian-Interventionist to optimize diet recommendations

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Body fat percent | Baseline, 12-months, 18-months
  The primary outcome is change from baseline body fat percent of the child at 12 or 18-month visit. Body fat percent is assessed by sum of the skin folds at 4 locations: triceps, thigh, subscapular, suprailiac.

SECONDARY OUTCOMES:
Body Mass Index (BMI) percentile | Baseline, 12-months, 18-months
  The secondary outcome is sex and age-specific BMI percentile of the child.

CONTACTS AND LOCATIONS:
Overall Officials: Linda V Van Horn, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Univeristy: Department of Preventive Medicine, Chicago, Illinois, United States